CLINICAL TRIAL: NCT01655277
Title: The Effects of Ultrasound Guided Adductor Canal Block Versus Femoral Nerve Block on Quadriceps Strength and Fall-risk: a Blinded Randomized Trial of Volunteers
Brief Title: Ultrasound Guided Adductor Canal Block Versus Femoral Nerve Block for Quadriceps Strength and Fall-risk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Principal Investigator, Jeff Gadsden, Director of Regional Anesthesia, St. Luke's-Roosevelt Hospital Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-202
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Quadriceps Muscle Weakness; Adductor Muscle Weakness; Fall Risk

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Adductor Canal block first (Experimental): This arm received an ultrasound guided adductor canal block with 15mL of chloroprocaine 3% followed by motor, sensory and balance assessments. Then the patients received an ultrasound guided femoral nerve block with 15mL of chloroprocaine 3% followed by sensory and motor assessments.
  Interventions: Procedure: Ultrasound Guided Adductor Canal Block; Procedure: Ultrasound Guided Femoral Nerve Block
- Femoral nerve block first (Experimental): This arm received an ultrasound guided femoral nerve block with 15mL of chloroprocaine 3% followed by motor, sensory and balance assessments. Then the patients received an ultrasound guided adductor canal block with 15mL of chloroprocaine 3% followed by sensory and motor assessments.
  Interventions: Procedure: Ultrasound Guided Adductor Canal Block; Procedure: Ultrasound Guided Femoral Nerve Block

INTERVENTIONS:
Procedure: Ultrasound Guided Adductor Canal Block
Procedure: Ultrasound Guided Femoral Nerve Block

SUMMARY:
Our objective was to determine if an ultrasound guided ACB can preserve quadriceps strength, thus minimizing weakness of knee extension compared with ultrasound guided femoral nerve block. Our primary outcome was the percent of maximum voluntary isometric contraction (MVIC) of knee extension preserved at 30 mins after either an ACB or FNB. Secondary outcomes included MVIC of knee extension at 60 min, hip adduction at 30 and 60 mins, and assessment of fall risk with the Berg Balance Scale (BBS) at 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18yrs)
* ASA 1-2

Exclusion Criteria:

* BMI >30
* Allergy to local anesthetics
* Pre-existing gait disturbance
* Pre-existing neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percent of maximum voluntary isometric contraction (MVIC) of knee extension preserved at 30 mins after either an ACB or FNB | At 30 minutes

SECONDARY OUTCOMES:
Percent of maximum voluntary isometric contraction (MVIC) of knee extension preserved at 60 mins after either an ACB or FNB | At 60 minutes
Percent of maximum voluntary isometric contraction (MVIC) of hip adduction preserved at 30 mins after either an ACB or FNB | At 30 minutes
Percent of maximum voluntary isometric contraction (MVIC) of hip adduction preserved at 60 mins after either an ACB or FNB | At 60 minutes
Assessment of fall risk with the Berg Balance Scale (BBS) at 30 minutes after the first nerve block. | At 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Roosevelt Hospital, New York, New York, United States